CLINICAL TRIAL: NCT04683432
Title: The Texture, Eating Rate and Glycaemic Index (TERAGI) Study
Acronym: TERAGI
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018/01091
Record Dates: First submitted 2020-12-16; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Adults
Keywords: Eating behaviour; Eating rate; Glycaemic response; Texture; Satiety
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: It is now recognized that diet plays a critical role in the etiology and management of chronic diseases such as type-2 diabetes, obesity and cardiovascular diseases. Evidence shows an increasing prevalence of type-2 diabetes as well as obesity, whereby large consumptions of carbohydrate foods is one of the leading contribution to these diseases. Food structure and texture can be modified to control oral processing behaviour, which would have subsequent impact on total energy intake and glycaemic response through altering the food breakdown path. Whilst it has been demonstrated that foods which are eaten at a faster rate leads to more food consumed ad-libitum and therefore higher energy intake, they are also eaten at fewer chews per bite, resulting in larger food particle sizes and hence slower digestion. Therefore it is important to understand the overall net effect of the opposing outcomes of food texture and oral processing behavior, bolus properties and glycaemic response, and identify the key factors which has the biggest influence on glycaemic response. The findings from this study can be used as guidelines on meal planning and making better informed choices between foods which are of the same composition/nutrition but with different health outcomes.

Study Aims: The aim of this study is to understand how food texture and saliva characteristics influences oral processing behavior, bolus characteristics and postprandial glycaemic response.

Study Design: Randomised crossover design where participants receive 2 treatments (i.e. 2 test meals) over 2 test sessions. Test sessions will include bolus characterisation of foods where participants chew and expectorate test foods (5g each) based on a fixed chew protocol.

Study Population: Up to 40 healthy males aged 21-50 years with BMI between 18-25 kg/m2

Intervention: For test session 1 and 2, participants will receive 2 treatments (i.e. 2 test meals) in randomised order over 2 sessions. The test meals contain 50g carbohydrate load of different textures. Participants will be video recorded while consuming the test meals to derive oral processing behaviour (bites, chews, time food spent in mouth). Blood samples will be collected at baseline and post consumption (5, 10, 15, 30, 45, 60, 90, 120 minutes) to measure glycaemic responses to the test meals. For test session 3, participants will be asked to follow a fixed chew protocol to chew and expectorate 3 test foods while being video recorded. Similarly, oral processing behaviours will be analysed from the recorded videos. The spat out food samples (i.e. bolus samples) will be analysed for saliva uptake and bolus particle size indicating extent of food breakdown.

DETAILED DESCRIPTION:
Study Aims:

The aim of this study is to understand how food texture and saliva characteristics influences oral processing behavior, bolus characteristics and postprandial glycaemic response.

The study hypothesizes that foods with a more elastic texture are eaten slower and requires more chewing, resulting in smaller bolus particle sizes and therefore higher postprandial glycaemic response due to an increased surface area for enzymatic digestion. Participants with higher saliva flowrate and/or alpha-amylase activity would also have shorter eating times and higher postprandial glycaemic responses.

Study Design:

Oral processing behaviours have high individual variances (Bolhuis et al 2013; Ketel et al 2019) and a large sample size is required in order to get significant differences between treatments. Based on previous papers on food texture and oral processing, a minimum of 20 healthy young male Chinese participants will be recruited in this study.

The study will require participants to attend 1 screening session (1 hour) and 3 test sessions (3 hours for test sessions 1 and 2; 1 hour for test session 3).

Screening (1 hour):

All potential participants will be asked to give informed consent before taking part in any of the research activities. Baseline measurements including anthropometric (height, weight, percentage body fat using a Bioelectrical Impedance Analyser), fasting blood glucose via finger prick and blood pressure will be taken to access eligibility.

Successfully screened participants will proceed to complete intraoral volume capacity measured using simple sip-and-spit measures, as well as provide stimulated and unstimulated saliva sample (approximately 4 x 5 ml each) via passive drooling to assess their saliva flowrates and saliva alpha-amylase activity.

Test Foods:

Commercially available and commonly consumed foods (e.g. white rice, korean rice cake, carrot, biscuits, etc.) are safe for human consumption and prepared in line with safe hygienic food preparation

Test session 1 and 2 (3 hours each):

Participants will be informed to fast 10 to 12 hours prior to test session 1 and 2. They are required to arrive the test centre between 08:00 - 09:00 a.m.

Participants will be asked to consume a test meal during each session, consisting of a 'fast' (less elastic texture and eaten more quickly) or 'slow' food (more elastic texture and eaten more slowly) in total. The order of test foods presented will be randomised. These test foods will be of the same carbohydrate load (50g carbohydrate) with different textures (i.e. white rice vs. rice cakes).

A baseline finger prick blood sample will be taken. After obtaining the baseline blood samples, test meal will be given to the participant to consumed within 15 minutes while being video recorded using a laptop webcam at face level. Following consumption of the test meal, finger prick blood samples will be taken for the next 5, 10, 15, 30, 45, 60, 90 and 120 minutes. The amount of blood that will be collected at every time point will be about a drop of blood (approximately 0.5ml per time point and 5 ml in total).

Sensory and textural ratings of the test meal will be taken using a visual analogue scale on a laptop. Post-meal satiety responses using a visual analogue scale will also be collected on a laptop every 15 minutes.

After completion of blood collection and satiety responses, the participant will be asked to chew on a separate portion of test meal (5g) until ready to swallow, and will be asked to expectorate the food bolus to assess their bolus properties including saliva uptake and particle size distribution. Video-recordings of the participant chewing the test foods will be taken.

A set of ad-libitum snacks will be provided to participants after all the measurements have been completed.

Test sessions 1 and 2 will be interspaced by a minimum of 5 days.

Test session 3 (1 hour):

Participants will be asked to chew on 3 test foods (white rice, rice cake, raw carrot) using a fixed chew protocol (i.e. 15 chews, 30 chews and chew until point of first swallow) and then expectorating the bolus to assess their bolus properties including saliva uptake and particle size distribution. Video-recordings of the participant chewing the test foods will be taken.

Sessions 2 and 3 will be interspaced by a minimum of 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese ethnicity
* Age between 21-40 years
* Weigh at least 45 kg
* Body mass index between 18to 25 kg/m²
* Normal blood pressure (</=140/90 mmHg)
* Fasting blood glucose <6.0 mmol/L
* Healthy dentition and ability to bite, chew and swallow normally
* No history of pain or discomfort in jaw movements or excessive teeth clenching or grinding, no caries or periodontal disease and no impaired salivation functions

Exclusion Criteria:

* Partake in sports at the competitive and/or endurance levels
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have known history of anaemia or thalassemia minor
* Have major chronic disease such as heart disease, cancer or diabetes mellitus
* Take insulin or drugs known to affect glucose metabolism
* Intentionally restrict food intake
* Have major medical or surgical event requiring hospitalization within the preceding 3 months
* Have taken antibiotics for 3 months before the study period
* Smoker
* Overnight shift worker
* Have any known food allergy (eg. anaphylaxis to peanuts)
* Have an active Tuberculosis (TB) condition or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus(HCV), Human Immunodeficiency Virus (HIV)
* Member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC
* Have poor veins impeding venous access
* Have any history of severe vasovagal syncope (blackouts or near faints) following blood draws

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males will be recruited. Hormonal fluctuations in females can affect glycaemic response.
Study Population: Males of Chinese ethnicity and aged between 21 to 40 years old.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Oral processing behaviour of test meal | During test session 1 (up to 3 hours)
  Participants will be video-recorded to measure oral processing behaviour of the test meal (white rice or rice cake)
Oral processing behaviour of test meal | During test session 2 (up to 3 hours)
  Participants will be video-recorded to measure oral processing behaviour of the test meals (white rice or rice cake)
Blood glucose response to test meal | During test session 1 (up to 3 hours)
  Blood glucose response will be measured through blood samples collected via finger prick at baseline (i.e. 0 minute) and post consumption of test meal (white rice or rice cake). (i.e. 0 min, 5 min, 10 min, 15 min, 30 min, 45 min, 60 min, 90 min and 120 min (0.5ml blood each)).
Blood glucose response to test meal | During test session 2 (up to 3 hours)
  Blood glucose response will be measured through blood samples collected via finger prick at baseline (i.e. 0 minute) and post consumption of test meal (white rice or rice cake). (i.e. 0 min, 5 min, 10 min, 15 min, 30 min, 45 min, 60 min, 90 min and 120 min (0.5ml blood each)).
Reported satiety in response to test meal | During test session 1 (up to 3 hours)
  Meal satiety responses using a visual analogue scale (VAS) will be collected on a laptop every 15 minutes during pre- and post- consumption of test meal (white rice or rice cake). VAS is anchored at 'Not at all full' (0) to 'Extremely full' (100), where a higher score will indicate greater satiety.
Reported satiety in response to test meal | During test session 2 (up to 3 hours)
  Meal satiety responses using a visual analogue scale (VAS) will be collected on a laptop every 15 minutes during pre- and post- consumption of test meal (white rice or rice cake). VAS is anchored at 'Not at all full' (0) to 'Extremely full' (100), where a higher score will indicate greater satiety.
Reported sensory and textural rating of test meal | During test session 1 (up to 3 hours)
  Meal satiety responses after test meal (white rice or rice cake) is consumed will be assessed using a visual analogue scale (VAS) will be collected on a laptop every 15 minutes during test session 1. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Reported sensory and textural rating of test meal | During test session 2 (up to 3 hours)
  Meal satiety responses after test meal (white rice or rice cake) is consumed will be assessed using a visual analogue scale (VAS) will be collected on a laptop every 15 minutes during test session 1. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Bolus characterisation of test meal | During test session 1 (up to 3 hours)
  Bolus characterisation of the test meal will be assessed by having participants chew a fixed mouthful of the test meal (white rice or rice cake, 5g) until ready to swallow, then expectorating it in a cup.
  Participants will be video-recorded to measure time and number of chews taken to swallow, before expectoration.
Bolus characterisation of test meal | During test session 2 (up to 3 hours)
  Bolus characterisation of the test meal will be assessed by having participants chew a fixed mouthful of the test meal (white rice or rice cake, 5g) until ready to swallow, then expectorating it in a cup.
  Participants will be video-recorded to measure time and number of chews taken to swallow, before expectoration.
Bolus characterisation of 3 test foods | During test session 3 (up to 1 hour)
  Bolus characterisation of the test meals will be assessed by having participants chew a fixed mouthful of the test foods (5g) based on a fixed chew protocol, then expectorating it in a cup.
  Participants will be video-recorded to measure time and number of chews taken to swallow, before expectoration.

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Forde, PhD, Principal Investigator — Ciaran_Forde@sifbi.a-star.edu.sg
Locations (1):
- Singapore Institute of Food and Biotechnology Innovation (SIFBI)/Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh AT, Chatonidi G, Choy M, Ponnalagu S, Stieger M, Forde CG. Impact of Individual Differences in Eating Rate on Oral Processing, Bolus Properties and Post-Meal Glucose Responses. Physiol Behav. 2021 Sep 1;238:113495. doi: 10.1016/j.physbeh.2021.113495. Epub 2021 Jun 9. PMID 34116051